CLINICAL TRIAL: NCT01409005
Title: A Phase II Trial of Gemcitabine Plus UFTE Combination Chemotherapy as Salvage Treatment in Oxaliplatin, Irinotecan and Fluoropyrimidine-Refractory Metastatic Colorectal Cancer
Brief Title: Gemcitabine-UFTE Chemotherapy in Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Seoul National University Hospital (Other); SMG-SNU Boramae Medical Center (Other); Yuhan Pharmaceutical Company (Unknown); Jeil Pharmaceutical Company (Unknown)
Responsible Party: Jee Hyun Kim, Department of Internal Medicine, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-SNU-2011-01
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic or Recurrent Colorectal Cancer; Refractory to Fluoropyrimidine, Oxaliplatin and Irinotecan; Salvage Chemotherapy
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine plus UFTE (Experimental): Gemcitabine plus UFTE chemotherapy (Single arm)
  Interventions: Drug: Gemcitabine and UFTE chemotherapy

INTERVENTIONS:
Drug: Gemcitabine and UFTE chemotherapy — Gemcitabine : 800 mg/m2 mix with 150mL of normal saline (i.v.) over 30 min on Days 1, 8 and 15
  UFTE : 200mg/m2 PO q 8 hr, Days 1~21
  Interval: every 4 weeks

SUMMARY:
Although there have been remarkable advances in the treatment of metastatic or recurrent colorectal cancer (MRCRC), long term survival cannot be expected in most patients with MRCRC because of inevitably developing resistance to chemotherapeutic drugs except some MRCRC patients who can undergo complete resection (metastasectomy). Until now, approved cytotoxic drugs for treatment of MCRC are only 3 categories (fluoropyrimidine, oxaliplatin and irinotecan). Recently, molecularly targeted drugs are approved for MRCRC patients, and bevacizumab and cetuximab (for K-ras wild type tumors) are available. When cytotoxic and targeted drugs are appropriately combined, about 24 months of overall survival (OS) can be expected in patients with MRCRC. However, when these drugs are all used or patients cannot afford to receive expensive targeted drugs because of economical problems, there is no option for chemotherapy and best supportive care is the only option, although some patients still have good performance status and medical conditions. Therefore, there are unmet needs for additional salvage chemotherapy regimens for patients with oxaliplatin, irinotecan and fluoropyrimidine-refractory MRCRC.

In some previous studies, gemcitabine-based chemotherapy showed some antitumor activities in MRCRC patients. Especially, when combined with fluoropyrimidine, gemcitabine has been shown to exert synergic effects on antitumor activities. On these backgrounds, this phase 2 clinical study was designed. In this study, efficacy and safety of gemcitabine plus UFTE chemotherapy will be evaluated in MRCRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* ECOG performance status: 0 to 2
* Pathologically proven adenocarcinoma of colorectum
* Patients who had received all cytotoxic drugs of 3 categories (fluoropyrimidine [5-FU, capecitabine or S-1 etc.], oxaliplatin and irinotecan).
* Refractory MRCRC that progressed while receiving, or within 6 months after the discontinuation of all of fluoropyrimidine, oxaliplatin and irinotecan. When retry of fluoropyrimidine, oxaliplatin or irinotecan is not possible due to previous severe toxicities despite progression-free interval ≥ 6 months, patients can be enrolled into this study.
* Patients who were previously treated with cetuximab or to whom cetuximab cannot be used (i.e. K-ras mutant or economical problems)
* At least one measurable lesion should exist (RECIST version 1.1)

Exclusion Criteria:

* Patients who had not previously received all of fluoropyrimidine, oxaliplatin and irinotecan will be excluded.
* Patients who had received UFTE chemotherapy previously. However, if UFTE chemotherapy was used as adjuvant chemotherapy and the disease-free interval was greater than 6 months, the patient can be included into this study.
* Patients receiving active or passive immunotherapy
* Patients with complete bowel obstruction or progressive symptoms of partial bowel obstruction that interfere with adequate oral diet.
* Patients with large amount of ascites requiring frequent therapeutic paracentesis (> once per week)
* Pregnant or breast-feeding women (a pregnancy test must be performed on all female patients who are of child-bearing potential before entering the study)
* Women of child-bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period. Sexually active fertile men not using effective birth control during the study if their partners are women of child-bearing potential
* Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy (i.e., uncontrolled infection, uncontrolled epilepsy, cerebrovascular accidents within the past 6 months, neurologic or psychological disease interfering with study treatment)
* Inadequate cardiovascular function:

  * New York Heart Association class III or IV heart disease,
  * Unstable angina or myocardial infarction within the past 6 months,
  * Symptomatic coronary artery disease
  * History of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
* Symptomatic severe interstitial lung disease or pulmonary fibrosis
* Patients with impaired renal function: Creatinine clearance < 50mL/min (calculated by Cockcroft and Gault formula)
* Patients with laboratory results as follows;

  * Number of absolute neutrophil counts (ANC) < 1.5 x 10^9/L
  * Number of thrombocytes < 100 x 10^9/L
  * Total bilirubin > 1.5 x upper limit of normal
  * ALAT, ASAT > 3 x upper limit of normal (in the cases with liver metastasis, > ALAT, ASAT > 5 x upper limit of normal)
  * Alkaline phosphatase > 3 x upper limit of normal (in the cases with liver or bone metastasis, > 5 x upper limit of normal)
* Major surgery within 4 weeks of start of study treatment, without complete recovery
* Patients who were included to other clinical trials within the past 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
8-weeks progression free survival rate (PFS rate) | Response evaluation using computed tomography (CT) at 8 weeks after the initiation of chemotherapy
  % of patients without tumor prgression at 8 weeks after the initiation of chemotherapy

SECONDARY OUTCOMES:
Overall survival (OS) | OS will be measured until death or study completion, with an expected average of 9 months
  OS will be measured until death of patients or study completion. Survival status will be followed up every 3 months if study treatment is completed.
Response rate (RR) | Response evaluation using CT will be performed every 8 weeks until tumor progression or death
  RECIST version 1.1 will be used for response evaluation
Percentage of Patients with Adverse Events | Overall safety will be monitored on every visit of patients during chemotherapy, with an expected average of 4 months
  Hematologic and non-hematologic toxicities will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Hyun Kim, M.D. & Ph.D., Principal Investigator — Professor, Department of Internal Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul
  - SMG-SNU Boramae Medical Center, Seoul, Seoul